CLINICAL TRIAL: NCT02533050
Title: Attentional Capacity and Working Memory in Coronary Artery Disease Patients: Impact of the Presence of a Sleep Apnea Syndrome and Chronic Effects of Treatment With a Continuous Positive Airway Pressure System (CPAP). Etude CAPCORSAS
Brief Title: Attentional Capacity and Working Memory in Coronary Artery Disease Patients: Impact of the Presence of a Sleep Apnea Syndrome and Chronic Effects of Treatment With CPAP
Acronym: CAPCORSAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1308171; 2013-A01635-40 (Other: ANSM)
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Apnea; Acute Coronary Syndrome
Keywords: obstructive sleep apnea; acute coronary event; cognitive functions; Continuous positive airway pressure night
MeSH Terms: conditions — Sleep Apnea, Obstructive; Acute Coronary Syndrome | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients treated (Experimental): Patients with CAD and SAS. This patients should have an apnea-hypopnea index (AHI) between 15 and 40, and an Epworth sleepiness score (ESS) <10. After randomization, they will be treated with CPAP treatment.
  Interventions: Device: CPAP treatment
- Patients non-treated (No Intervention): Patients with CAD and SAS. This patients should have an apnea-hypopnea index (AHI) between 15 and 40, and an ESS <10. After randomization, they will be not treated.
- Control group (No Intervention): Patients with CAD but without SAS (AHI<15).

INTERVENTIONS:
Device: CPAP treatment — Patients treated wear a face mask during sleep which is connected to a pump (CPAP machine) that forces air into the nasal passages at pressures high enough to overcome obstructions in the airway and stimulate normal breathing.
  Arms: Patients treated

SUMMARY:
The presence of Obstructive Sleep Apnea Syndrome (OSAS) has a high frequency in patients victims of a coronary artery disease (CAD) (myocardial infarction, revascularization). Unlike patients seen in a sleep Laboratory with an impact on daytime functioning, CAD apneic patients do not complain in their daytime functioning. The objective of this study is to explore whether the objective cognitive assessment measures may be a good marker of the efficacy of CPAP treatment given to non-sleepy apneic CAD patients.

Coronary patients with an AHI between 15 and 40 / h will be treated (or not) after randomization with CPAP treatment. The expected results are: CPAP apneic coronary patients should have a positive impact on cognitive performance, particularly on attention span and working memory measured by improvement in the Paced Auditory Serial Addition Test score (PASAT score).

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the Clinical Physiology Department of Exercise of the Saint Etienne University Hospital (myocardial infarction, coronary stenting or coronary artery bypass) and referred for care in cardiac rehabilitation
* A native French speaker
* No daytime sleepiness (ESS <or = 10)
* Signature of informed consent by the patient

Exclusion Criteria:

* Patients with a previous diagnosis of sleep apnea syndrome
* Patients with severe heart failure (stage III and IV of the NYHA)
* Patients with a neurodegenerative disease or other known cognitive disorders
* Presence of progressive disease other than coronary artery disease (cancer for example)
* Patients participating in other research that can change their cognitive function or drowsiness

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-02-24 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
PASAT-4sec test score | Day 120
  The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. Single digits are presented every 4 seconds and the patient must add each new digit to the one immediately prior to it. The score for the PASAT is the total number correct out of 60 possible answers.

SECONDARY OUTCOMES:
Score Mini Mental State (MMS) | Day 120
  It is a score obtained in psychometric tests. This is a series of 30 questions that assesses cognitive and mnemonic ability of a person.
Mean time (ms) obtained in a Continus Performance Test | Day 120
  It is an other score obtained in psychometric tests. It measures a person's sustained and selective attention (associated with impulsivity and distractibility).
Percentage (%) obtained in a test measurement of the reaction time | Day 120
  It is an other score obtained in psychometric tests. It is a psychometer vigilance test.
Mean time (ms) obtained in a test measurement of the reaction time | Day 120
  It is an other score obtained in psychometric tests. It is a psychometer vigilance test.
Percentage (%) for a N-back working memory task | Day 120
  It is an other score obtained in psychometric tests. The subject is presented with a sequence of stimuli, and the task consists of indicating when the current stimulus matches the one from n steps earlier in the sequence.
Average time (ms) for a N-back working memory task | Day 120
  It is an other score obtained in psychometric tests. The subject is presented with a sequence of stimuli, and the task consists of indicating when the current stimulus matches the one from n steps earlier in the sequence.
AHI | Day 120
  It is the number of apnea and hypopnea per hour. It determined by polysomnography.
Mean nocturnal oxygen saturation (%) | Day 120
  It is a percentage index of hypoxemia measured by a polysomnography.
Minimal nocturnal oxygen saturation (%) | Day 120
  It is an other percentage index of hypoxemia measured by a polysomnography.
The oxyhemoglobin desaturation index | Day 120
  It is an other index of hypoxemia measured by a polysomnography. It is expressed in desaturations / hour
The time (min) spent with a SaO2 below 90% | Day 120
  The arterial oxygen saturation (SaO2)is an other index of hypoxemia measured by a polysomnography.
Sleep fragmentation | Day 120
  It is determined by a polysomnography.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic ROCHE, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No